CLINICAL TRIAL: NCT00571571
Title: Application and Evaluation of Transference Focused Psychotherapy Modified for Adolescents
Acronym: TFP-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Anna E. Odom, Ph.D., Weill Cornell Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0610008834
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Identity Pathology; Behavior Problems
Keywords: Identity difussion; Adolescent psychotherapy; Transference Focused Psychotherapy for Adolescents; Identity; Identity crisis; Identity pathology
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TFP-A (Experimental): Specific aspects of TFP-A involve the setting up of a treatment contract/collaboration between patient and therapist to deal with the likely threats both to the treatment and to the patient's well being that may occur in the course of the treatment. After the behavioral symptoms of identity pathology are contained through structure and limit setting, the psychological structure that is believed to be the core of identity pathology are analyzed. In particular, treatment would involve the family in setting up the contract parameters, provide a psychoeducational component to the family and patient, inclusion of school personnel as appropriate to reinforce contract parameters, place an emphasis on the technique of clarification to understand specific emotional states.
  Interventions: Behavioral: Psychotherapy
- Control (Active Comparator): The Control Group is treatment as usual in the outpatient clinic. Treatment in this arm will be carried out by therapists in the Outpatient Department. Treatment will be determined by the therapist(s) and carried out according to their particular orientation and their assessment of patient's needs. It is expected based on clinic data that the majority of patients will be seen at least one time per week.
  Interventions: Behavioral: Individual Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Individual psychotherapy with parent collateral/psychoeducation as necessary.
  Other Names: TFP-A; Transference Focused Psychotherapy for Adolescents
  Arms: TFP-A
Behavioral: Individual Psychotherapy — Individual psychotherapy and family interventions (as needed)
  Arms: Control

SUMMARY:
Normal adolescence requires a successful resolution of identity crisis, which results in the development of satisfying relationships, success in school/work pursuits, and achievement of personal goals. Adolescents, who do not resolve this crisis, are at high risk for problems in those areas of functioning. Transference Focused Psychotherapy for Adolescents (TFP-A) is a treatment that specifically addresses these issues, permitting adolescents to develop satisfying friendships, more appropriate interactions with authority, and achieve realistic life goals.

This study will evaluate the application of TFP-A, (a empirically validated treatment for adults with identity disturbance), to adolescents exhibiting the same behavioral and identity pathology. Subjects will be females; ages 14-21, with behaviors associated with identity problems, interpersonal difficulties with teachers, parents and/or peers, and live with their families. These adolescents will be randomly assigned to one of two treatment cells, TFP-A or Treatment as Usual (TAU). Subjects in TFP-A will receive weekly individual therapy for six months. The TAU group will receive standard individual therapy in the Outpatient Department. Both will receive medication as necessary. All subjects will participate in initial, weekly, and bi-monthly assessments during the six-month treatment period, and participate in a naturalistic follow-up study for an additional six months.

Hypothesis:

Adolescents with identity problems as seen in interpersonal, school, and/or family difficulties in the Transference Focused Psychotherapy for Adolescents (TFP-A) group will reduce these problem behaviors and improve management of their feelings and moods compared to adolescents with identity problems in the treatment as usual control group (TAU).

ELIGIBILITY:
Inclusion Criteria:

1. Female Adolescents, ages 14-21
2. A score of five out of nine critical items on the Borderline Personality Disorder Dimension Interview Scale.
3. Have interpersonal difficulties in school, family, and/or peer functioning.
4. Live at home with family.
5. Willingness to attend evaluation sessions and weekly, individual therapy.

Exclusion Criteria:

1. The presence of psychosis, substance dependence, non-verbal learning disability, antisocial behavior, and/or primary diagnoses of eating disorder, bipolar disorder, and obsessive-compulsive disorder.
2. The need for hospitalization for symptom management.
3. Significant cognitive impairment (Full Scale IQ <85).
4. The presence of a life-threatening medical illness.

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in interpersonal difficulties with parents, teachers, and/or peers. Improved management of their feelings and moods. Reduction in other problems behaviors (i.e. substance use, self-injurious behaviors) | Subjects will be assessed at entry, 2 month, 4 months, 6 months, 8 months 10 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Odom, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York-Presbyterian Hospital, White Plains, New York, United States

REFERENCES:
- [Background] Clarkin JF, Foelsch PA, Levy KN, Hull JW, Delaney JC, Kernberg OF. The development of a psychodynamic treatment for patients with borderline personality disorder: a preliminary study of behavioral change. J Pers Disord. 2001 Dec;15(6):487-95. doi: 10.1521/pedi.15.6.487.19190. PMID 11778390
- [Background] Clarkin JF, Levy KN, Lenzenweger MF, Kernberg OF. Evaluating three treatments for borderline personality disorder: a multiwave study. Am J Psychiatry. 2007 Jun;164(6):922-8. doi: 10.1176/ajp.2007.164.6.922. PMID 17541052
- [Background] Clarkin JF, Levy KN, Lenzenweger MF, Kernberg OF. The Personality Disorders Institute/Borderline Personality Disorder Research Foundation randomized control trial for borderline personality disorder: rationale, methods, and patient characteristics. J Pers Disord. 2004 Feb;18(1):52-72. doi: 10.1521/pedi.18.1.52.32769. PMID 15061344